CLINICAL TRIAL: NCT05079204
Title: Effectiveness of Intraoral Scanners as a Motivation Method for Oral Hygiene Instruction
Brief Title: Intraoral Scanners as a Motivation Method for Oral Hygiene Instruction
Acronym: Perio3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PO20159*
Record Dates: First submitted 2021-10-05; First posted 2021-10-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis; Gingivitis
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator which perform the periodontal examination will be blinded of the motivation procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional motivation procedure (Active Comparator): Conventional motivation procedures defined as a presentation of the modified Bass technique on a dental teaching macro model plus intra oral instruction provided in patient's mouth with a hand mirror.
  Interventions: Other: No intervention
- Conventional motivation procedure supported by 3D representations (Experimental): Conventional motivation procedures associated with 3D intra oral procedures. A 3D intra-oral modelization will added to the previously described procedure. Then, a periodontist will show the sites contaminated by dental plaque to the patient.
  Interventions: Other: Intra oral scan

INTERVENTIONS:
Other: Intra oral scan — Cover key details of the intervention. Must be sufficiently detailed to distinguish between arms of a study and/or among similar interventions Intervention consists in an 3D intra oral representation of the oral cavity.
  Other Names: Conventional motivation procedures supported by 3D representations
  Arms: Conventional motivation procedure supported by 3D representations
Other: No intervention — No intervention
  Arms: Conventional motivation procedure

SUMMARY:
Periodontal diseases are highly prevalent inflammatory diseases. These diseases are mostly due to the development and the maturation of bacterial plaque which lead to local inflammation. Individuals can develop severe attachment loss which could lead to dental loss. To prevent them, individual plaque removal procedures self-performed by the patient by tooth brushing or interdental brushes or made by professional care (scaling), are known to improve periodontal health, and thus to prevent periodontal diseases. Moreover, oral hygiene is a major factor to increase increasing the outcomes when treatments are needed. However, patients' compliance in oral health program is one of the major limits to periodontal therapeutics.

In this study, the investigators evaluate the effectiveness of 3D intra-oral camera compared with conventional oral hygiene instructions, to improve oral health motivation.

DETAILED DESCRIPTION:
The present study explores the effectiveness of intraoral scanners in the field of oral hygiene motivation and instruction to improve the patient's motivation.

Patients presenting periodontitis or gingivitis are recruited and randomized in 2 groups: conventional motivation procedures and conventional motivation procedures supported with 3D representations of their mouth obtained by intraoral scanners. Periodontal diseases (periodontitis and gingivitis) will be diagnosed according to the international classification of periodontal diseases, based on the decision-making algorithms. A periodontal charting, socio-demographic data and clinical data will be collected. Then, oral mucosa dermatological manifestations, treatment needs (ICDAS) and quality of life related to oral health (GOHAI) will be evaluated.

After inclusion, patients will be randomized between conventional motivation procedures and conventional motivation procedures associated with 3D intra oral procedures.

The investigators hypothesized that the 3D intra oral representations could improve oral hygiene in patients compared with those receiving only a classical motivation procedure. The primary objective is to evaluate if patients instructed to oral hygiene procedures using a representation of their mouth obtained by the use of a intraoral scanner present fewer plaque than the ones instructed without it. This could be achieved by the analysis of plaque control record index in both group.

The secondary objectives are :

* To compare the evolution of the bleeding on probing clinical index between the two groups.
* To compare the evolution of mean periodontal pocket depths, mean recessions and mean clinical attachment level between the two groups.
* To compare the quality of life related to oral health between the two groups
* To evaluate the time needed to add intraoral scans in the procedure
* To evaluate the relevance of the received information.

ELIGIBILITY:
Inclusion Criteria:

Patients

* consulting the Dental Care Service of the university hospital of Reims
* presenting gingivitis or periodontal diseases according to the international classification of periodontal diseases (Chicago, 2017)
* presenting at least 10 pairs of opposing teeth
* able to perform oral hygiene procedures
* speaking French
* who signed the informed consent form
* affiliated to the French Social Security system

Non-inclusion criteria :

Patients presenting :

* a medical history likely to compromise protocol (psychiatric disorders, medical or pharmacological antecedents altering or modifying immune response in last 3 months)
* pregnancy or breastfeeding
* eating disorders
* orthodontic treatments
* patients under legal protection, trusteeship or guardianship
* unable to understand auto-questionary

Exclusion criteria :

Patients presenting :

* presenting exacerbations signs of periodontal diseases
* benefiting a professional plaque removal procedure outside of the experimental procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Plaque Control Record Evolution | Day 14
  Recording the presence of plaque on individual tooth surfaces (mesial, distal, facial, lingual). The plaque is highlighted by a periodontal probe.
  PCR is calculated according the following formula :
  PCR = (Number of faces with plaque / Total number of faces) x 100

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: No